CLINICAL TRIAL: NCT03871933
Title: Characterization of Autonomic Function in Patients With Chronic Obstructive Pulmonary Disease - Potential Relevance for Increased Risk of Atrial Fibrillation
Brief Title: Autonomic Function in COPD and Risk for Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Principle Investigator, Heinrich-Heine University, Duesseldorf
Other Study IDs: 16-029
Record Dates: First submitted 2019-03-11; First posted 2019-03-12 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: atrial fibrillation; autonomic function; cardiopulmonary interaction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collection of 20 ml of peripheral blood Clinical routine such as NTproBNP, renal function, thyroid function, blood count
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AECOPD: acute exacerbation of COPD
  Interventions: Other: Measurement of lung function, electrocardiography, echocardiography and autonomic function
- stable COPD
  Interventions: Other: Measurement of lung function, electrocardiography, echocardiography and autonomic function

INTERVENTIONS:
Other: Measurement of lung function, electrocardiography, echocardiography and autonomic function — Measurement of lung function, electrocardiography, echocardiography and autonomic function

SUMMARY:
In the presented study, autonomic function as well as risk for atrial fibrillation will be assessed to characterize the relation between risk of atrial fibrillation and autonomic function.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) has been suggested as relevant comorbidity in patients with chronic obstructive pulmonary disease (COPD). The evaluation of the total atrial conduction time via tissue Doppler imaging (PA-TDI interval) can be used to identify patients with increased risk of new onset AF. Autonomic function can be assessed by different non invasive clinical investigations.

The investigators hypothesise that PA-TDI interval is increased in acutely exacerbated COPD (AECOPD) compared within stable COPD and that increased PA-TDI is related to impairment of autonomic function. For this purpose, 25 patients with AECOPD and 25 patients with stable COPD were characterized by clinical characteristics, laboratory tests, lung function, electrocardiography, echocardiography and autonomic function.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic obstructive pulmonary disease, exacerbated or stable between the age of 40-80 years with sinus rhythm who gave informed written consent

Exclusion Criteria:

* Inability to give written consent, acute myocardial infarction with ST-segment elevations in last 30 days, severe acute or chronic renal dysfunction, severe heart failure, atrial fibrillation, severe valve disease, severe hypotension, active malignant disease, active rheumatic disease

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic obstructive pulmonary disease, exacerbated or stable
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
total atrial conduction time | Baseline
  total atrial conduction time via tissue Doppler imaging (PA-TDI interval)

SECONDARY OUTCOMES:
Heart rate variability | Baseline
  For the assessment of autonomic function different test that characterize sympathetic or parasympathic function are performed. All tests for autonomic function are non invasive.
Baroreflex sensitivity | Baseline
  For the assessment of autonomic function different test that characterize sympathetic or parasympathic function are performed. All tests for autonomic function are non invasive.
Chemoreflex sensitivity | Baseline
  For the assessment of autonomic function different test that characterize sympathetic or parasympathic function are performed. All tests for autonomic function are non invasive.
Deep breathing test | Baseline
  For the assessment of autonomic function different test that characterize sympathetic or parasympathic function are performed. All tests for autonomic function are non invasive.
Ewing test | Baseline
  For the assessment of autonomic function different test that characterize sympathetic or parasympathic function are performed. All tests for autonomic function are non invasive.
Cold pressure test | Baseline
  For the assessment of autonomic function different test that characterize sympathetic or parasympathic function are performed. All tests for autonomic function are non invasive.
Cold face test | Baseline
  For the assessment of autonomic function different test that characterize sympathetic or parasympathic function are performed. All tests for autonomic function are non invasive.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Düsseldorf, Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No